CLINICAL TRIAL: NCT01044966
Title: Phase I/II Intraventricular DepoCyt (OD # 06-2348) in Glioblastoma (76,730, 11/06)
Brief Title: A Study of Intraventricular Liposomal Encapsulated Ara-C (DepoCyt) in Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of adequate patient enrollment into trial.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3542; R01FD003542-01 (FDA); NCT01026168 (obsolete NCT alias)
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma Multiforme; Glioma; Astrocytoma; Brain Tumor
Keywords: Glioblastoma; Subventricular; gliomagenesis; temozolomide; depocyt
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITV DepoCyt + Temozolomide (Experimental): Patients will undergo an induction phase of intraventricular (ITV) DepoCyt, using the dosage determined from the Phase I portionPatients with stable disease (clinically and radiographically), not exhibiting systemic toxicity, will undergo a three month consolidation phase of ITV DepoCyt, for one month (Cycles 3-6). Patients without progression or toxicity will undergo maintenance therapy using ITV DepoCyt every four weeks (+/- 3 days) for a maximum of 8 months (cycles 7-14) or until recurrence or toxicity ensues. Oral metronomic Temozolomide dosing of 75 mg/m2 daily for 21 days followed by 7 days off will be given throughout the Induction, Consolidation, and Maintenance Phases of the ITV DepoCyt described above.
  Interventions: Drug: ITV DepoCyt + Temozolomide

INTERVENTIONS:
Drug: ITV DepoCyt + Temozolomide — Intrathecal liposomal Ara-C dosing will begin at 50 mg ITV every 2-4 weeks, and de-escalated based on toxicity obtained from the Phase I portion of the trial. Metronomic dosing of temozolomide will be given at 75 mg/m2 for 21 days (continuous oral dosing), followed by 7 days off in a 28 day cycle as a once daily dosing regimen.
  Other Names: Intrathecal liposomal Ara-C (DepoCyt); Temozolomide (Temodar)

SUMMARY:
Current treatments for Glioblastoma Multiforme (GBM), the most common and malignant primary brain tumor are inadequate and as such, the median survival for most patients with GBM is on the order of months, even after cytoreductive surgery, radiation and chemotherapy. This study aims to develop a new treatment for GBM by suppressing glial progenitor cells that surround the ventricular system in patients with these aggressive tumors because it is these regions that appear to act as an incubator for future recurrences resulting in patient death. Considering the lack of significant treatment options for patients with this uniformly fatal disease, this is an important translational clinical study to perform.

DETAILED DESCRIPTION:
Despite significant improvements in diagnostic imaging and neurosurgical techniques, the current treatment modalities for high-grade gliomas are inadequate. As such, the median survival for most patients with GBM is on the order of months, even after cytoreductive surgery, radiation and chemotherapy. Fewer than 3% of GBM patients are still alive at 5 years after diagnosis. A rising incidence has been reported for GBM, and the survival rate for patients with GBM has not shown improvement in the last two decades. For this reason exploring novel therapies for the treatment of GBM is warranted.

Neuro-oncology is currently in the midst of a paradigm shift in terms of our accepted understanding of the pathophysiology of gliomagenesis. Classic "dedifferentiation" hypotheses, modeling the cellular origin of gliomas after neoplastic transformation of differentiated glia, are currently being challenged by hypotheses suggesting dysregulated glial progenitor cells are responsible for gliomagenesis. Growing evidence exists that glial progenitor cells persisting in the adult mammalian brain, lining the lateral ventricles in the subventricular zone (SVZ) and dentate gyrus, play a role in gliomagenesis. Gliomas frequently occur in close proximity to the ventricular system and SVZ with high-grade lesions like GBM "spreading" to midline structures and crossing the corpus callosum to the contralateral hemisphere. Glial progenitor cells lining the lateral ventricles in the SVZ and dentate gyrus may be the source of "tumor" cells "spreading" to midline structures such as the corpus callosum as well as continuously replenishing the tumor bed resulting in local recurrences.

The lack of significant clinical advances in treating GBM may be due to oversight of the SVZ component of this disease. It is our hypothesis that successful treatment of GBM will require suppression of the SVZ component in addition to the currently accepted modalities of hemispheric tumor resection followed by radiation and chemotherapy. This understanding of gliomagenesis has not yet been used clinically for the treatment of GBM. We hypothesize that the SVZ is the incubator for future recurrences of GBM and propose targeting SVZ progenitor cells with intraventricular liposomal encapsulated Ara-C (DepoCyt) in combination with systemic metronomic dose temozolomide. Ara-C has been previously demonstrated to inhibit the proliferation and migration of SVZ precursor cells in adult animals. Two patients treated using this novel regimen have demonstrated significant responses warranting further study of this treatment in the Phase I/II clinical trial proposed here. This has also been the basis for successful application and granting of Orphan-Drug designation for cytarabine (Ara-C) liposome injection (trade name: DepoCyt) for the treatment of gliomas (Designation # 06-2348) on January 30, 2007.

ELIGIBILITY:
Inclusion Criteria:

* Age Patients must be at least 18 years of age but no older than 85 years.
* Diagnosis Patients with the histological diagnosis of recurrent GBM made either by biopsy or resection of recurrent disease. Cytological evidence of malignant cells in CSF and/or clinical and radiographic evidence of leptomeningeal disease are irrelevant in terms of inclusion or exclusion into this study. Bihemispheric extension ("butterfly GBM"), multi-focality, and/or subependymal spread are not contraindications to enrollment.
* Prior therapy Patients must have had an initial diagnosis of "malignant glioma" (WHO grade III or IV) and failed initial surgical resection followed by standard adjuvant therapy including external beam radiotherapy to a 2cm margin of 60 Gy, and standard temozolomide chemotherapy of 150 to 200 mg per square meter for 5 days during each 28-day cycle prior to "recurrence." Patients must not have received more than one other systemic or ITV adjuvant chemotherapy regimen in addition to temozolomide prior to enrollment, not including intracavitary Gliadel wafer placement. Prior Gliadel wafer placement is not a contradiction to patient enrollment in this trial.
* Performance Status Patients must have Karnofsky performance status (KPS) of ≥ 60%.
* Recovery from Prior Therapy Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy, prior to entering this study and must be without significant systemic illness (e.g. infection unresponsive to treatment after 7 days). Such that they are healthy enough to safely undergo tumor biopsy and Ommaya reservoir placement. Patients must not have received any systemic therapy for recurrent disease within 3 weeks (6 weeks if a nitrosourea), or irradiation within 8 weeks prior to treatment on this study.
* Hematologic Status Patients must have a platelet count > 75,000/mm3 and ANC > 1500/mm3 within 72 hours prior to ITV DepoCyt treatment.
* Hepatic and Renal Status Patients must have adequate liver function (total bilirubin < 2.0 mg%; ALT, and AST < 4 times normal); adequate renal function (serum creatinine <1.6 mg, and BUN < 22); normal serum electrolytes (sodium, potassium, calcium, magnesium, and phosphorus).
* Informed Consent (See Appendix) All patients or their legal guardians must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study.

Exclusion Criteria:

* Patients younger than 18 or older than 85 years of age.
* Patients with histological diagnoses other than recurrent GBM.
* Patients with a Karnofsky performance status (KPS) < 60%.
* Patients that have received more than one other systemic or ITV adjuvant chemotherapy regimen in addition to temozolomide, not including intracavitary Gliadel wafer placement.
* Patients concurrently receiving other therapies (either brachytherapy or systemic) designed specifically to treat the recurrent GBM.
* Patients within 8 weeks of receiving stereotactic or external beam irradiation.
* Patients with a platelet count < 75,000/mm3 and ANC < 1500/mm3 within 72 hours prior to ITV DepoCyt and/or oral temozolomide treatment.
* Patients with liver dysfunction (total bilirubin > 2.0 mg%; ALT, and AST > 4 times normal).
* Patients with renal dysfunction (serum creatinine >1.6 mg, and BUN > 22).
* Patients with abnormal serum electrolytes (sodium, potassium, calcium, magnesium, and phosphorus).
* Patients with contraindications to having placement of a ventricular access device such as Ommaya reservoir.
* Patients with clinical and/or neuroradiographic evidence of hydrocephalus or increased intracranial pressure.
* Patients with signs and symptoms of systemic infection precluding them from receiving chemotherapy or prohibiting Ommaya reservoir placement.
* Pregnant and breast feeding women will be excluded. All other women of childbearing years must have a negative serum pregnancy test.
* Patients with a ventricular-peritoneal or ventricular-atrial shunt.
* Prisoners will be excluded from this study.
* Patients or their legal guardians not willing or able to sign the informed consent document.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Frankel, MD, Principal Investigator — Medical University of South Carolina, Dept. of Neurosciences, Division of Neurosurgery; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- See also: (Link to contact Dr. Frankel at Medical University of South Carolina) — http://www.muschealth.com/findadoc?Action=DoctorInfo&Doctor_ID=2365&gclid=CNGXpYyeuZ4CFQ...

RESULTS

PARTICIPANT FLOW:
Groups:
- ITV DepoCyt + Temozolomide: Patients will undergo an induction phase of intraventricular (ITV) DepoCyt, using the dosage determined from the Phase I portionPatients with stable disease (clinically and radiographically), not exhibiting systemic toxicity, will undergo a three month consolidation phase of ITV DepoCyt, for one month (Cycles 3-6). Patients without progression or toxicity will undergo maintenance therapy using ITV DepoCyt every four weeks (+/- 3 days) for a maximum of 8 months (cycles 7-14) or until recurrence or toxicity ensues.
  ITV DepoCyt + Temozolomide: Intrathecal liposomal Ara-C dosing will begin at 50 mg ITV every 2-4 weeks, and de-escalated based on toxicity obtained from the Phase I portion of the trial. Metronomic dosing of temozolomide will be given at 75 mg/m2 for 21 days (continuous ora
Period: Induction Phase
Arm/Group | ITV DepoCyt + Temozolomide
Started | 12
Completed | 12
Not Completed | 0
Period: Consolidation Phase
Arm/Group | ITV DepoCyt + Temozolomide
Started | 12
Completed | 2
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.9 [32 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: The type and number of adverse events will be recorded and reported by the number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- ITV DepoCyt + Temozolomide: Patients will undergo an induction phase of intraventricular (ITV) DepoCyt, using the dosage determined from the Phase I portionPatients with stable disease (clinically and radiographically), not exhibiting systemic toxicity, will undergo a three month consolidation phase of ITV DepoCyt, for one month (Cycles 3-6). Patients without progression or toxicity will undergo maintenance therapy using ITV DepoCyt every four weeks (+/- 3 days) for a maximum of 8 months (cycles 7-14) or until recurrence or toxicity ensues.
  ITV DepoCyt + Temozolomide: Intrathecal liposomal Ara-C dosing will begin at 50 mg ITV every 2-4 weeks, and de-escalated based on toxicity obtained from the Phase I portion of the trial. Metronomic dosing of temozolomide will be given at 75 mg/m2 for 21 days (continuous oral dosing), followed by 7 days off in a 28 day cycle as a once daily dosing regimen.
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: Proportion of Patients With Recurrent GBM Treated With ITV DepoCyt in Combination With Oral Temozolomide Who Are Progression-free at 16 Weeks.
Description: Eligibility of patients with GBM that are able to receive study drug to estimate the proportion of patients with recurrent GBM treated with ITV DepoCyt in combination with oral temozolomide who are progression-free at 16 weeks. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Progression Free Survival
Description: The progression free survival of patients receiving study drug will be recorded. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Response Rate of Drug Treatment
Description: Those responding to study drug will be recorded. Response will be defined as stable neurological examination in conjunction with the absence of progression as defined above.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Participants | 2

5. Secondary Outcome: Quality of Life Outcomes Measurement
Description: Participants recorded are those who had an improvement in QOL score, QOL outcomes will be assessed and recorded using the EORTC QLQ C30 version 3.
  This 30 question questionnaire will be used to asses our patient overall feeling of well-being during the trial. Questions to assess quality of life are measured from 1-4 with the following graded values:
  1. Not at all
  2. A little
  3. Quite a bit
  4. Very much Lower total scores are consistent with better quality of life and changes of greater or equal to 10 points are considered a significant change in quality of life.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ITV DepoCyt + Temozolomide
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Arm/Group | ITV DepoCyt + Temozolomide
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITV DepoCyt + Temozolomide (N=12)
CSF leak (Surgical and medical procedures) | 1 (1) — Leak from Ommaya
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITV DepoCyt + Temozolomide (N=12)
seizure (Nervous system disorders) | 1 (1) — Patients with seizures after treatment administered

LIMITATIONS AND CAVEATS:
The enrollment of patients in this study was limited due to a number of factors including: rareness of disease, poor KPS upon disease recurrence, the availability of subsequent FDA approved drugs (Avastin) after study initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No